CLINICAL TRIAL: NCT02924623
Title: Discordance Dans l'évaluation d'Activité de la Polyarthrite Rhumatoide
Brief Title: Discrepancies Between Patients and Physicians in Their Perceptions of Rheumatoid Arthritis Disease Activity
Acronym: DIAPO
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: LOCAL/2015/CGV-03
Record Dates: First submitted 2016-09-16; First posted 2016-10-05 (Estimated); Last update posted 2019-04-25 (Actual); Status verified 2019-01

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional

SUMMARY:
Patients and physicians often differ in their perceptions of rheumatoid arthritis (RA) disease activity, as quantified by the patient's global assessment (PGA) and by the evaluator's global assessment (EGA).

The objectives of this study were:

1. to explore the extent and reasons for the discordance between patients and physicians in their perception of RA disease activity
2. to determine if this discordance at baseline is associated with RA outcomes at 1 year (remission, function and structure) in early arthritis (EA) in daily clinical practice.

   * Patients: from the French cohort of early arthritis (EA) ESPOIR³ (at least 2 swollen joints for less than 6 months, DMARD naïve), fulfilling the ACR-EULAR criteria for RA at baseline

Analysis: At baseline, agreement between PGA and EGA (Bland-Altman plot) was assessed. Multivariate linear regression was used to determine the patient and EA features independently associated with discordance (calculated as PGA - EGA). Logistic regression was used to analyze discordance as│PGA - EGA│≥20.

Multivariate logistic models were used to determine if discordance at baseline is associated with remissions (Boolean, SDAI and DAS28), functional stability (HAQ≤0.5 and deltaHAQ≤0.25) and absence of radiographic progression (delta Sharp score<1) after 1 year of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* fulfilling the ACR-EULAR criteria for RA

Exclusion Criteria:

* no RA

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: from the south of France (Nîmes, Montpellier, Toulouse, Bordeaux, Limoge), fulfilling the ACR-EULAR criteria for RA
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
Patient's global assessment | day 0
  The discordance between the patient's and the evaluator's global assessment will be calculated.
Evaluator's global assessment | day 0
  The discordance between the patient's and the evaluator's global assessment will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Cécile Gaujoux-Viala, MD, PhD, Principal Investigator — CHU Nîmes
Locations (1):
- CHU Nîmes, Nîmes, Gard, France